CLINICAL TRIAL: NCT07023419
Title: Psychiatric Disorders in Addiction - Interest of Screening and Influence on Relapse
Acronym: Psyaddict
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9533
Record Dates: First submitted 2025-03-24; First posted 2025-06-17 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-03

CONDITIONS: Psychiatric Disorders
Keywords: Psychiatric Disorders; Addiction; Complex detox
MeSH Terms: conditions — Mental Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In complex detoxification hospital units, patients receive a common care system (interviews, therapeutic workshops, support for discharges, etc.). In the event of a relapse during hospitalization, i.e., a relapse into addiction, hospital care is called into question, and discharge is generally considered. A key care issue is therefore to prevent these relapses by identifying risk profiles to strengthen their management. According to studies, psychiatric diagnoses increase the risk of relapse, but the investigators do not fully understand which ones or to what extent.

The objective of this study is to analyze the influence of psychiatric diagnoses on the risk of relapse. This would allow for adapting the care of these patients to reduce this risk. The investigators are also seeking to study the value of screening questionnaires in improving the reliability of psychiatric diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged ≥16
* Having been hospitalized in the complex withdrawal unit of the Strasbourg psychiatric clinic during the period from January 1, 2024 to November 1, 2024

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subject aged ≥16 and having been hospitalized in the complex withdrawal unit of the Strasbourg psychiatric clinic during the period from January 1, 2024 to November 1, 2024
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Score (ISI) | At 22 months
  The ISI is a scale composed of 7 questions:
  Each of the 7 items is rated on a 5-point Likert scale (from 0 to 4). The total score is obtained by adding the scores for all 7 items (1a+1b+1c+2+3+4+5). The total score ranges from 0 to 28:
  0-7 = No insomnia 8-14 = Subclinical (mild) insomnia 15-21 = Clinical (moderate) insomnia 22-28 = Clinical (severe) insomnia
Depression Scale Score (PHQ 9) | At 22 months
  Depression Scale Score (PHQ 9)
  * Items are rated on a scale from 0 to 3. The maximum score is 27.
  * The threshold for assessing moderate depression (10 or higher) is the most commonly used. • Thresholds:
  No depression: 0-4 points; Mild depression: 5-9 points; Moderate depression: 10-14 points; Moderately severe depression: 15-19 points; Severe depression: 20-27 points.
Anxiety score (GAD-7) | At 22 months
  Anxiety score (GAD-7):
  The total score of the GAD-7 questionnaire ranges from 0 to 21 points. Scores of 5, 10, and 15 represent thresholds for detecting mild, moderate, or severe anxiety:
  Score 0-4: Minimal anxiety Score 5-9: Mild anxiety Score 10-14: Moderate anxiety Score above 15: Severe anxiety
Posttraumatic Stress Disorder Score (PCL-5) | At 22 months
  Posttraumatic Stress Disorder Score (PCL-5):
  The PCL-5 scale assesses the presence and severity of PTSD using 20 items.
  The PTSD severity score ranges from 0 (not present at all) to 4 (extremely), resulting in a total score between 0 and 80. PCL-5 scores were used to determine the presence of PTSD.:
  A score:
  above 33 indicates the presence of PTSD, between 31 and 33 indicates probable PTSD below 31 indicates no PTSD.
Addictions Score (DAST-10) | At 22 months
  Addictions Score (DAST-10):
  The maximum total score is 10. A threshold of 3 or 4 is recommended for screening for a drug use problem. This threshold would most closely match the criteria in the Diagnostic and Statistical Manual of Mental Disorders (DSM):
  A score of 9 or higher indicates a severe problem.
ADHD Score | At 22 months
  ADHD Score:
  Points are summed on a scale of 0 to 24, with a threshold of 14 or higher for a positive ADHD screen result. The total score can be categorized into four strata:
  0 to 9 = weakly negative 10 to 13 = strongly negative 14 to 17 = weakly positive 18 to 24 = strongly positive
Autism Score (RAADS-14) | At 22 months
  Autism Score (RAADS-14):
  The RAADS-R test calculates a score indicating the likelihood of an autism spectrum disorder in the individual taking it. The total score on the RAADS-R test ranges from 0 to 240.
  Higher scores indicate behaviors and symptoms consistent with autism. Scores equal to or greater than 65 indicate the presence of autism.
Emotion Dysregulation Score (DERS-16) | At 22 months
  Emotion Dysregulation Score (DERS-16) A 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: (1) cognitive reappraisal and (2) expressive suppression. Respondents respond to each item on a 7-point Likert-type scale, ranging from 1 (strongly disagree) to 7 (strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Addictologie - CHU de Strasbourg - France, Strasbourg, France